CLINICAL TRIAL: NCT06222281
Title: Evaluation of Shoulder Strength and Deltoid Stiffness After RSA
Brief Title: Evaluation of Shoulder Strength and Deltoid Stiffness After Reverse Shoulder Arthroplasty (RSA)
Status: Completed | Type: Observational
Sponsor: Şensu Dinçer (Other)
Responsible Party: Sponsor-Investigator, Şensu Dinçer, medical doctor, Istanbul University
Organization: Istanbul University (Other)
Other Study IDs: Elastography RSA
Record Dates: First submitted 2024-01-04; First posted 2024-01-24 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Sonoelastography; Isokinetic Test
Keywords: elastography; Deltoid; shoulder strength; reverse shoulder arthroplasty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to test the strength of the shoulder joint and elasticity of the deltoid muscle of the patients who had a reverse shoulder arthroplasty. The main questions are: • Whether there is a difference between the operated and healthy shoulders in terms of strength and deltoid elasticity of the patients. • Is there any correlation between the functional status, elasticity and strength of the operated shoulder? Participants will be asked to attend the isokinetic shoulder strength tests and shear wawe ultrasound elastography measurements. They will be also asked to fill the quick DASH and Constant score forms.

DETAILED DESCRIPTION:
The ultrasound elastography is a measurement method that has become increasingly common recently and can measure some mechanical properties of tissue. Measurements can be made using two different techniques: strain and shear wave elastography (SWEUS). SWEUS provides objective and reproducible data collection about the elasticity of the tissue and is less affected by the user than the strain technique. The mechanical properties of the deltoid muscle are among the main factors affecting surgical results in patients undergoing reverse shoulder replacement surgery. Glenohumeral joint function is affected by the post-operative tension of the deltoid. Excessive tension in the deltoid muscle may cause restriction of movement and pain, as well as conditions such as instability and insufficient force production. Lack of elasticity of deltoid muscle may also lead to functional deficit of shoulder. Previous studies have found a linear correlation between muscle activity and muscle elasticity values measured by MR elastography (MRE). However, MRE is an expensive method that requires large equipment and space, and it is a more difficult method for patients, which may include various difficulties in patient positioning. Ultrasound elastography is a method that is highly investigated for clinical use because it is cheaper and easier to apply than MRE. Isokinetic dynamometer is one of the most objective methods used to measure muscle activity and strength.Thus, it is imperative to reveal the mechanical properties of deltoid muscle, which carries the most of the mechanical load in the shoulder region after the operation, as well as the relationship between them.

The medical history of patients who had undergone reverse prosthesis surgery in the Department of Orthopedics and Traumatology, and their postoperative files will be screened. Patients who meet the inclusion and exclusion criteria will be invited to the study.

Their demographic information will be recorded. The visual pain scale (VAS) and will be questioned to evaluate the pain status. Functional status of the patients, and the patients will be asked to complete the Constant score and the quick arm, shoulder and hand problems questionnaire (Q-DASH) under supervision. They will be asked to answer. Shear wave elastographic measurement and isokinetic tests of both shoulders will be carried out in the sports medicine department. Measurement outcomes of both shoulders will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Having undergone reverse shoulder arthroplasty surgery due to arthropathy because of unilateral rotator cuff tear
* Followed for at least 12 months after surgery.
* The other unoperated shoulder is healthy.

Exclusion Criteria:

* Patients with revision reverse shoulder arthroplasty
* Having inflammatory diseases
* Not having adequate range of motion to be able to perform isokinetic test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were operated in the university hospital, department of orthopedics and traumatology
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
shear wave elastography (SWE) | Through study completion, an average of 8 weeks
  SWE provides an indirect measure of a tissue's mechanical properties by quantifying the speed at which sound waves propagate through soft tissue. Shear wave elastography will be carried out once for both shoulders before the isokinetic tests
shoulder adduction strength | Through study completion, an average of 8 weeks
  adduction strength of both shoulders will be measured by the isokinetic test method. It will be carried out once for both shoulders for each patient. To measure the muscle strength, the average peak torque (nm) done with four repetitions at a velocity of 60 /sec was determined. It will be carried out once for both shoulders for each patient. Results will be presented in newton metre (nm) unit
shoulder adduction endurance | Through study completion, an average of 8 weeks
  endurance strength of both shoulders will be measured by the isokinetic test method. It will be carried out once for both shoulders for each patient. To measure the muscle strength, the average peak torque (nm) done with four repetitions at a velocity of 180 /sec was determined. It will be carried out once for both shoulders for each patient. Results will be presented in newton metre (nm) unit.
modified Constant shoulder outcome score | It will be carried out once for each patient, through study completion, an average of 8 weeks
  Patients will fill the constant score questionnaire to evaluate the functional status of operated shoulder. The modified Constant score will be used to determine the functionality after the treatment of a shoulder injury. The test is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points).The higher the score, the higher the quality of the function
American Shoulder Elbow Surgeons (ASES) orthopedic score | It will be carried out once for each patient, through study completion, an average of 8 weeks
  The ASES is a condition-specific scale that is intended to measure functional limitations and pain of the shoulder.
Quick shoulder disabilities arm shoulder and hand questionnaire (QuickDASH) | It will be carried out once for each patient, through study completion, an average of 8 weeks
  Patients will fill the quick disabilities of the arm, shoulder, and hand outcome measure questionnaire (the quick-DASH) to evaluate the functional status of operated shoulder.his questionnaire is a self-report questionnaire that patients can rate difficulty and interference with daily life on a 5 point Likert scale.t is a questionnaire that measures an individual's ability to complete tasks, absorb forces, and severity of symptoms.The QuickDASH tool uses a 5-point Likert scale from which the patient can select an appropriate number corresponding to his/her severity/function level.
shoulder abduction endurance | Through study completion, an average of 8 weeks
  to measure the shoulder abduction endurance, total work (nm) done with 15 repetitions at a velocity of 180/sec will be measured by an isokinetic dynamometer, results will be presented in newton metre (nm) unit
shoulder abduction strength | Through study completion, an average of 8 weeks
  adduction strength of both shoulders will be measured by the isokinetic test method. It will be carried out once for both shoulders for each patient. To measure the muscle strength, the average peak torque (nm) done with four repetitions at a velocity of 60 /sec was determined. It will be carried out once for both shoulders for each patient. Results will be presented in newton metre (nm) unit

CONTACTS AND LOCATIONS:
Locations (1):
- Şensu Dinçer, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No